CLINICAL TRIAL: NCT01957293
Title: Influence of Salbutamol on Emotional and Cognitive Functions in Healthy Subjects
Acronym: Salmon-Basel
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Prof. Dominique de Quervain, MD (Other)
Collaborators: Clinical Trial Unit, University Hospital Basel, Switzerland (Other)
Responsible Party: Sponsor-Investigator, Prof. Dominique de Quervain, MD, Director of teh Division of Cognitive Neuroscience, University of Basel
Organization: University of Basel (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 2013DR2134
Record Dates: First submitted 2013-09-24; First posted 2013-10-08 (Estimated); Last update posted 2014-12-16 (Estimated); Status verified 2014-02

CONDITIONS: Memory Functions
MeSH Terms: interventions — Albuterol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Salbutamol (Experimental)
  Interventions: Drug: Salbutamol
- Sugar Syrup (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Salbutamol — single oral administration, 4 mg
  Arms: Salbutamol
Drug: Placebo — single oral administration
  Arms: Sugar Syrup

SUMMARY:
Aim is to investigate the effect of beta2 adrenergic stimulant salbutamol on emotional and cognitive functions in healthy humans.

ELIGIBILITY:
Inclusion Criteria:

Healthy, male and female, aged between 18 and 40, BMI be-tween 19 and 27 kg/m2, normotensive (BP between 90/60 mmHg and 140/90 mmHg), native or fluent German-speaking, caucasian (European ancestry), able and willing to give written informed consent and comply with the requirements of the study protocol, willing to donate saliva sample for DNA-analysis -

Exclusion Criteria:

Acute or chronic psychiatric or somatic disorder, tachycardia at rest (> 100 bpm), known hypersensitivity to salbutamol, pathological ECG, pregnancy, breast-feeding, long-term medication within last 3 months (oral contraceptives are disregarded) smoking (>3 cigarettes per day), concurrent participation in another study, participation in one of our previous studies using the same memory tests, inability to read and understand the participant's information. -

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2013-10; Primary Completion 2014-01 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Change of emotional memory functions under Salbutamol | two testing days within 10 days
  memory tests
Change of episodic memory functions under Salbutamol | two testing days within10 days
  memory tests

SECONDARY OUTCOMES:
Change of emotional state under salbutamol | Two testing days within 10 days
  questionnaires
change of attention functions under salbutamol | two testing days within 10 days
  attention tests

CONTACTS AND LOCATIONS:
Overall Officials: Dominique de Quervain, Prof. MD, Study Director — University of Basel
Locations (1):
- University of Basel, Division of Cognitive neuroscience, Basel, Switzerland